CLINICAL TRIAL: NCT06939504
Title: Evaluation of the Relative Bioavailability of HRS-9813 Capsule and Tablet in Healthy Subjects and the Effect of Food on the Pharmacokinetics of HRS-9813 Capsule
Brief Title: A Trial of HRS-9813 Capsule and Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HRS-9813-103
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-9813 Capsule Group (Experimental)
  Interventions: Drug: HRS-9813 Capsule
- HRS-9813 Tablet Group (Experimental)
  Interventions: Drug: HRS-9813 Tablet

INTERVENTIONS:
Drug: HRS-9813 Capsule — HRS-9813 capsule.
  Arms: HRS-9813 Capsule Group
Drug: HRS-9813 Tablet — HRS-9813 tablet.
  Arms: HRS-9813 Tablet Group

SUMMARY:
This is a phase Ⅰ study to evaluate the relative bioavailability of HRS-9813 capsule and tablet in healthy subjects and the effect of food on the pharmacokinetics of HRS-9813 capsule.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-45 years.
2. Male weight ≥ 50 kg, female weight ≥ 45 kg, and body mass index (BMI): 19-26 kg/m2.
3. Subjects not with clinically significant vital signs and laboratory tests.
4. Take contraception measures.

Exclusion Criteria:

1. Any serious clinical diseases that affect the absorption, metabolism and/or excretion of the study drug.
2. Severe infection, severe trauma or major surgery.
3. Any medications in the two weeks before screening or baseline period.
4. History of blood donation or severe blood loss.
5. Have been vaccinated within 2 weeks before the screening or baseline period.
6. History of smoking or excessive alcohol or drug abuse.
7. Other situations that the researcher judges to be unsuitable.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-05-04 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration of HRS-9813 capsule (Cmax) | Day 1-Day 23.
Maximum observed concentration of HRS-9813 tablet (Cmax) | Day 1-Day 23.
Area under the concentration-time curve from time 0 to infinity of HRS-9813 tablet (AUC0-inf) | Day 1-Day 23.
Area under the concentration-time curve from time 0 to infinity of HRS-9813 capsule (AUC0-inf) | Day 1-Day 23.

SECONDARY OUTCOMES:
Adverse events (AEs) | Day 1-Day 23.
Time to Cmax of HRS-9813 capsule (Tmax). | Day 1-Day 23.
Time to Cmax of HRS-9813 tablet (Tmax). | Day 1-Day 23.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided